CLINICAL TRIAL: NCT03915834
Title: Biomarkers to Predict Hemorrhage and Outcomes After Endovascular Treatment in Patients With Acute Large Vessel Occlusion
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Other Study IDs: 2018-033
Record Dates: First submitted 2019-03-18; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Acute Ischemic Stroke
Keywords: Biomarker; Mechanical thrombectomy; Intracerebral Hemorrhage; Acute Ischemic stroke
MeSH Terms: conditions — Ischemic Stroke; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- endovascular treatment group
  Interventions: Device: Endovascular treatment

INTERVENTIONS:
Device: Endovascular treatment — Mechanical thrombectomy and/or Aspiration

SUMMARY:
The main aim of the biomarkers to predict Hemorrhagic transformation(HT) after endovascular treatment in Acute Ischemic Stroke Patients.

The study has three main parts. During the first part, the investigators propose to conduct an enrollment of patients after thrombectomy in acute Ischemic Stroke and healthy controls. Serum biomarkers levels were analyzed (before and after) endovascular treatment patients and controls respectively.

During the second part, HT was evaluated and classified on cranial computed tomography and/or MRI post- treatment and was considered as symptomatic HT (sHT) if associated with neurological deterioration.

During the third part, the investigators aim to demonstrate the level of biomarkers can significant predict HT and outcomes in stroke patients undergoing revascularization.

ELIGIBILITY:
Inclusion Criteria:

1. be 18 or older;
2. have a clinical diagnosis of acute ischemic stroke
3. a score of 6 or more points on the NIHSS(the National Institutes of Health Stroke Scale);
4. be scheduled to undergo intraarterial (IA) therapy for acute hemispheric stroke;
5. patients eligible for IV alteplase should receive IV alteplase;
6. Intracranial arterial occlusion of the distal intracranial carotid artery, middle (M1/M2) ,anterior (A1/A2) cerebral artery,vertebral artery,basilar artery or posterior cerebral artery,demonstrated with CTA, MRA or DSA;
7. begin intra-arterial therapy within 24 hours of symptom onset;
8. have provided informed consent.

Exclusion Criteria:

1. have any pre-existing illness resulting in a modified Rankin Scale Score of 3 or higher prior to the qualifying stroke;
2. patients with known infectious, inflammatory, or neoplastic diseases at the time of treatment and non-availability of blood samples;
3. are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke patients
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-04-16 (Estimated); Primary Completion 2019-10-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Hemorrhagic transformation | 24 to 72 hours
  Hemorrhagic transformation was diagnosed by Computed tomographic scans usually performed 24 to 72 hours after the procedure.Symptomatic intracranial hemorrhage was defined as neurologic deterioration (an increase of 4 or more points in the score on the NIHSS) and evidence of intracranial hemorrhage on imaging studies.

SECONDARY OUTCOMES:
Modified Rankin scale | 90 days
  this scale measures functional outcome, with scores ranging from 0 (no symptoms) to 6 (death).scores of the modified Rankin scale at 2 years (0 or 1 [excel- lent outcome], 0 to 2 [good outcome, indicating functional independence], and 0 to 3 [favorable outcome]).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xuan Wu Hospital，Capital Medical University, Beijing, Beijing Municipality
  - Beijing Luhe Hospital, Capital Medical University, Beijing